CLINICAL TRIAL: NCT00772486
Title: A Phase 1b Study of Repeated Doses of Autologous CLL B Cells Transduced to Express Chimeric CD154 (ISF35) in Combination With Fludarabine, Cyclophosphamide and Rituximab (FCR) in Subjects With Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Phase Ib Study of ISF35 in Combination With Chemotherapy (FCR) in Subjects With Relapsed, Refractory, and/or 17p- CLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memgen, LLC (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Organization: Memgen, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL-35-104; NCT00796016 (obsolete NCT alias)
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2010-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Immune System Diseases; Rituximab; Fludarabine; Cyclophosphamide; ISF35; Ad-ISF35; Refractory; Resistant; 17p-; del 17p; 17p; Resistant CLL; Refractory CLL; 17p- CLL; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Leukemia, B-Cell; Immune System Diseases; Chromosome 17 deletion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: ISF35 and FCR (Experimental): ISF35 and FCR
  Interventions: Biological: ISF35

INTERVENTIONS:
Biological: ISF35 — Subjects participating in this study will receive a course of three infusions of 3x10^8 ISF35-transduced cells at periods of not less than 14 days apart followed by a standard regimen of three cycles of fludarabine, cyclophosphamide and rituximab (FCR) at monthly intervals.
  Other Names: Ad-ISF35; AdISF35

SUMMARY:
The study is a Phase 1b open label, non-randomized, single institution clinical trial that is designed to evaluate the safety and tolerability of three repeat infusions of ISF35 followed by a standard regimen of three cycles of fludarabine, cyclophosphamide and rituximab (FCR) in subjects with refractory, resistant, and/or 17p- CLL.

DETAILED DESCRIPTION:
ISF35 has already been used in two Phase I clinical trials. The trials demonstrated that ISF35 treatment is well tolerated and patients did not experience any significant or unexpected adverse events. Patients reported flu-like symptoms from ISF35, which disappeared within one to three days.

The trials also showed that ISF35 stimulates the immune system to act against CLL cells and sensitize leukemic cells to subsequent treatment. Repeat infusions of ISF35 administered as a single agent to subjects with CLL resulted in durable reductions in circulating and lymph-node bound leukemic cells. Furthermore, CLL patients with 17p deletion responded to standard courses of FCR after receiving ISF35 and achieved durable remissions.

ISF35 is an abbreviation for Immune Stimulatory Factor 35, an offspring of technology discovered by Dr. Thomas J. Kipps, MD, PhD, Professor, Department of Medicine and Deputy Director for Research,UCSD Moores Cancer Center.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must have a diagnosis of B cell CLL including:

   * Lymphocytosis of monoclonal B-cells co-expressing ≥ one B-cell marker (CD19, CD20, or CD23) and CD5 in peripheral blood or lymph node AND
   * Bone marrow with ≥ 30% mononuclear cells having the CLL/SLL phenotype
2. Measurable disease, and at least one of the IWCLL 2008 Guidelines "Indications for Treatment" as follows:

   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia.
   * Massive (i.e., >6 cm below the left costal margin) or progressive or asymptomatic splenomegaly.
   * Massive nodes (i.e., >10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.
   * Progressive lymphocytosis with an increase of >50% over a 2-month period, or lymphocyte doubling time (LDT) of less than 6 months. LDT can be obtained by linear regression extrapolation of absolute lymphocyte counts (ALC) obtained at intervals of two weeks over an observation period of 2-3 months; patients with initial blood lymphocyte counts of less than 30,000 per microliter may require a longer observation period to determine the LDT. Also, factors contributing to lymphocytosis or lymphadenopathy other than CLL (e.g, infections) should be excluded.
   * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroids or other standard therapy.
   * A minimum of any one of the following disease-related symptoms must be present:
   * Unintentional weight loss ≥10% within the previous 6 months.
   * Significant fatigue (i.e., ECOG PS 2 or worse; cannot work or unable to perform usual activities).
   * Fevers of greater than 100.5 degrees F or 38.0 degrees C for 2 or more weeks without other evidence of infection.
   * Night sweats for more than 1 month without evidence of infection. Hypogammaglobulinemia or monoclonal or oligoclonal paraproteinemia does not by itself constitute a basis to initiate treatment.
3. Subjects must have CLL that is documented to be resistant or refractory to standard chemotherapy regimens containing alkylating agents and/or purine analogues. Chemotherapy refractory or resistant is defined as the following:

   * CLL progression during treatment (2 cycles) with chemotherapy; OR
   * Failure to achieve a PR or CR after at least 2 cycles of chemotherapy; OR
   * No response to treatment or stable disease after at least 2 cycles of chemotherapy; OR
   * Disease progression within 6 months of treatment with chemotherapy; OR
   * CLL with cytogenetic changes documenting the loss of the short arm of chromosome 17 (17p-) associated with the loss of p53.
4. Subjects must be age 18 years or older
5. For men and women of child-bearing potential, use of effective barrier contraceptive methods during the study and for one month following treatment
6. Subjects must have ECOG performance scale of ≤ 2
7. Subjects must have adequate hematologic, renal, hepatic, and coagulation function defined as:

   • Adequate hematologic function:

   i) Platelet count ≥ 50,000/µL; AND

   ii) Hemoglobin ≥ 10 g/dL (may be supported by erythropoietin or transfusion); AND

   • Adequate renal function:

   i) Calculated creatinine clearance ≥ 30 mL/min/1.73 m^2; OR

   ii) Serum creatinine ≤ 2 times upper limit of normal; AND

   • Adequate hepatic function:

   i) Total bilirubin ≤ 2.5 times upper limit of normal; AND

   ii) ALT ≤ 2.5 times upper limit of normal; AND

   • Adequate coagulation tests:

   i) Prothrombin time international normalized ratio (INR) ≤ 1.5; AND

   ii) Partial thromboplastin time ≤ 1.5 times upper limit of normal
8. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments

Exclusion Criteria

1. Presence of > 55% prolymphocytes or Richter's transformation
2. Chemotherapy (e.g., purine analogues, alkylating agents, or corticosteroids), antibody therapy, immunotherapy, radiation therapy, or participation in any investigational drug treatment within 4 weeks of enrollment into protocol or at any time during the study
3. Ongoing toxicity from prior anti-neoplastic therapy
4. Untreated autoimmune hemolytic anemia or immune thrombocytopenia
5. Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral (A, B or C) hepatitis
6. Positive serologies for HIV1,2 or HTLV I,II
7. CMV disease with positive DNA PCR
8. Syphilis with positive VDRL
9. Acute Hepatitis A and C with positive serologies, and Hepatitis B, acutely or chronically infected based on CDC criteria
10. Any illness or condition that in opinion of the investigator may affect safety of treatment or evaluation of any study's endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Assess toxicity, tolerability, and safety of repeat administration of three infusions of 3x10^8 ISF35 given intravenously in combination with a standard course of three treatments of fludarabine, rituximab and cyclophosphamide (FCR). | Duration of the Trial

SECONDARY OUTCOMES:
Explore the anti-leukemia activity of the repeat administration of ISF35 and FCR by evaluating reduction in leukemia count, reduction in lymphadenopathy and splenomegaly, improvement in bone marrow function, and response duration. | Duration of the Trial
Assess induction of B and T cell anti-leukemia immune responses, antibody production against autologous CLL B cells, changes in bystander leukemia cell phenotype, and expression of genes and proteins related to apoptosis | Duration of the Trial

CONTACTS AND LOCATIONS:
Overall Officials: Januario Castro, MD, Principal Investigator — Assistant Clinical Professor in the Blood and Marrow Transplantation Division
Locations (1):
- University of California, San Diego Moores Cancer Center, San Diego, California, United States

REFERENCES:
- [Background] Keating MJ, O'Brien S, Albitar M, Lerner S, Plunkett W, Giles F, Andreeff M, Cortes J, Faderl S, Thomas D, Koller C, Wierda W, Detry MA, Lynn A, Kantarjian H. Early results of a chemoimmunotherapy regimen of fludarabine, cyclophosphamide, and rituximab as initial therapy for chronic lymphocytic leukemia. J Clin Oncol. 2005 Jun 20;23(18):4079-88. doi: 10.1200/JCO.2005.12.051. Epub 2005 Mar 14. PMID 15767648
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Rai KR. Characteristics and Management of Chronic Lymphocytic Leukemia. Advances in Oncology. 1996;9 No.1:17-20.
- [Background] Kalil N, Cheson BD. Chronic lymphocytic leukemia. Oncologist. 1999;4(5):352-69. PMID 10551552
- [Background] Kay NE, Hamblin TJ, Jelinek DF, Dewald GW, Byrd JC, Farag S, Lucas M, Lin T. Chronic lymphocytic leukemia. Hematology Am Soc Hematol Educ Program. 2002:193-213. doi: 10.1182/asheducation-2002.1.193. PMID 12446424
- [Background] Bosch F, Montserrat E. Refining prognostic factors in chronic lymphocytic leukemia. Rev Clin Exp Hematol. 2002 Dec;6(4):335-49; discussion 449-50. doi: 10.1046/j.1468-0734.2002.00302.x. No abstract available. PMID 12823776
- [Background] Byrd JC, Waselenko JK, Keating M, Rai K, Grever MR. Novel therapies for chronic lymphocytic leukemia in the 21st century. Semin Oncol. 2000 Oct;27(5):587-97. PMID 11049025
- [Background] Nabhan C, Gartenhaus RB, Tallman MS. Purine nucleoside analogues and combination therapies in B-cell chronic lymphocytic leukemia: dawn of a new era. Leuk Res. 2004 May;28(5):429-42. doi: 10.1016/j.leukres.2003.08.017. PMID 15068894
- [Background] Nabhan C, Dyer MJ, Rosen ST. Current status of monoclonal antibody therapy for chronic lymphocytic leukemia. Oncology (Williston Park). 2003 Feb;17(2):253-62; discussion 264, 267, passim. PMID 12632866
- [Background] Byrd JC, Stilgenbauer S, Flinn IW. Chronic lymphocytic leukemia. Hematology Am Soc Hematol Educ Program. 2004:163-83. doi: 10.1182/asheducation-2004.1.163. PMID 15561682
- [Background] Rozman C, Montserrat E. Chronic lymphocytic leukemia. N Engl J Med. 1995 Oct 19;333(16):1052-7. doi: 10.1056/NEJM199510193331606. No abstract available. PMID 7675049
- [Background] Ghia P, Caligaris-Cappio F. The origin of B-cell chronic lymphocytic leukemia. Semin Oncol. 2006 Apr;33(2):150-6. doi: 10.1053/j.seminoncol.2006.01.009. PMID 16616061
- [Background] Chiorazzi N, Rai KR, Ferrarini M. Chronic lymphocytic leukemia. N Engl J Med. 2005 Feb 24;352(8):804-15. doi: 10.1056/NEJMra041720. No abstract available. PMID 15728813
- [Background] Perz J, Topaly J, Fruehauf S, Hensel M, Ho AD. Level of CD 20-expression and efficacy of rituximab treatment in patients with resistant or relapsing B-cell prolymphocytic leukemia and B-cell chronic lymphocytic leukemia. Leuk Lymphoma. 2002 Jan;43(1):149-51. doi: 10.1080/10428190210178. PMID 11908720
- [Background] Cheson BD, Bennett JM, Rai KR, Grever MR, Kay NE, Schiffer CA, Oken MM, Keating MJ, Boldt DH, Kempin SJ, et al. Guidelines for clinical protocols for chronic lymphocytic leukemia: recommendations of the National Cancer Institute-sponsored working group. Am J Hematol. 1988 Nov;29(3):152-63. doi: 10.1002/ajh.2830290307. PMID 3189311
- [Background] Lin TS, Lucas MS, Byrd JC. Rituximab in B-cell chronic lymphocytic leukemia. Semin Oncol. 2003 Aug;30(4):483-92. doi: 10.1016/s0093-7754(03)00239-2. PMID 12939717
- [Background] O'Brien SM, Kantarjian H, Thomas DA, Giles FJ, Freireich EJ, Cortes J, Lerner S, Keating MJ. Rituximab dose-escalation trial in chronic lymphocytic leukemia. J Clin Oncol. 2001 Apr 15;19(8):2165-70. doi: 10.1200/JCO.2001.19.8.2165. PMID 11304768
- [Background] Byrd JC, Rai K, Peterson BL, Appelbaum FR, Morrison VA, Kolitz JE, Shepherd L, Hines JD, Schiffer CA, Larson RA. Addition of rituximab to fludarabine may prolong progression-free survival and overall survival in patients with previously untreated chronic lymphocytic leukemia: an updated retrospective comparative analysis of CALGB 9712 and CALGB 9011. Blood. 2005 Jan 1;105(1):49-53. doi: 10.1182/blood-2004-03-0796. Epub 2004 May 11. PMID 15138165
- [Background] Wierda W, O'Brien S, Wen S, Faderl S, Garcia-Manero G, Thomas D, Do KA, Cortes J, Koller C, Beran M, Ferrajoli A, Giles F, Lerner S, Albitar M, Kantarjian H, Keating M. Chemoimmunotherapy with fludarabine, cyclophosphamide, and rituximab for relapsed and refractory chronic lymphocytic leukemia. J Clin Oncol. 2005 Jun 20;23(18):4070-8. doi: 10.1200/JCO.2005.12.516. Epub 2005 Mar 14. PMID 15767647
- [Background] Kipps TJ. Chronic lymphocytic leukemia and related diseases. In: Beutler E, Lichtman MA, Coller BS, Kipps TJ, Seligsohn U, eds. Williams Hematology (ed 6). New York: McGraw-Hill, Inc.; 2001:1163-1194.
- [Background] Wierda WG, Cantwell MJ, Woods SJ, Rassenti LZ, Prussak CE, Kipps TJ. CD40-ligand (CD154) gene therapy for chronic lymphocytic leukemia. Blood. 2000 Nov 1;96(9):2917-24. PMID 11049967
- [Background] Dicker F, Kater AP, Fukuda T, Kipps TJ. Fas-ligand (CD178) and TRAIL synergistically induce apoptosis of CD40-activated chronic lymphocytic leukemia B cells. Blood. 2005 Apr 15;105(8):3193-8. doi: 10.1182/blood-2003-10-3684. Epub 2004 Aug 31. PMID 15339846
- [Background] Chu P, Deforce D, Pedersen IM, Kim Y, Kitada S, Reed JC, Kipps TJ. Latent sensitivity to Fas-mediated apoptosis after CD40 ligation may explain activity of CD154 gene therapy in chronic lymphocytic leukemia. Proc Natl Acad Sci U S A. 2002 Mar 19;99(6):3854-9. doi: 10.1073/pnas.022604399. Epub 2002 Mar 12. PMID 11891278
- [Background] Dohner H, Stilgenbauer S, Benner A, Leupolt E, Krober A, Bullinger L, Dohner K, Bentz M, Lichter P. Genomic aberrations and survival in chronic lymphocytic leukemia. N Engl J Med. 2000 Dec 28;343(26):1910-6. doi: 10.1056/NEJM200012283432602. PMID 11136261
- [Background] Cantwell MJ, Sharma S, Friedmann T, Kipps TJ. Adenovirus vector infection of chronic lymphocytic leukemia B cells. Blood. 1996 Dec 15;88(12):4676-83. PMID 8977261
- See also: LLS, Memgen Collaborate on CLL Clinical Trial — http://www.leukemia-lymphoma.org/all_news_detail?item_id=520809&cat_id=140